CLINICAL TRIAL: NCT05798520
Title: A 2-Part, Multicenter, Randomized, Blinded, Active-Controlled Phase 2 Study to Sequentially Evaluate the Safety and Efficacy of BIIB091 Monotherapy and BIIB091 Combination Therapy With Diroximel Fumarate in Participants With Relapsing Forms of Multiple Sclerosis
Brief Title: A Study to Learn About the Safety of BIIB091 and Its Effect on Brain Inflammation When Taken Alone or With Diroximel Fumarate (DRF) in Adults With Relapsing Forms of Multiple Sclerosis (MS)
Acronym: FUSION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 257MS201; 2022-502552-31 (Other: EU CT NUMBER)
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: Multiple Sclerosis; Diroximel fumarate; BIIB091
MeSH Terms: conditions — Multiple Sclerosis | interventions — BIIB091

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: BIIB091 High Dose + Matching Placebo for DRF (Experimental): Participants will receive BIIB091 high dose and matching placebo for DRF, orally, for up to 48 weeks.
  Interventions: Drug: BIIB091; Drug: Placebo
- Part 1: BIIB091 Low Dose + Matching Placebo for DRF (Experimental): Participants will receive BIIB091 low dose and matching placebo for DRF, orally, for up to 48 weeks.
  Interventions: Drug: BIIB091; Drug: Placebo
- Part 1: DRF + Matching Placebo for BIIB091 (Active Comparator): Participants will receive DRF standard dose and matching placebo for BIIB091, orally, for up to 48 weeks.
  Interventions: Drug: DRF; Drug: Placebo
- Part 2: BIIB091 + DRF Standard Dose (Experimental): Participants will receive selected dose of BIIB091 (based on Part 1 data) and DRF standard dose, orally, for up to 48 weeks.
  Interventions: Drug: BIIB091; Drug: DRF
- Part 2: BIIB091 + DRF Low Dose (Experimental): Participants will receive selected dose of BIIB091 (based on Part 1 data) and DRF low dose, orally, for up to 48 weeks.
  Interventions: Drug: BIIB091; Drug: DRF
- Part 2: DRF + Matching Placebo for BIIB091 (Active Comparator): Participants will receive DRF standard dose and matching placebo for BIIB091, orally, for up to 48 weeks.
  Interventions: Drug: DRF; Drug: Placebo

INTERVENTIONS:
Drug: BIIB091 — Administered as specified in the treatment arm.
  Arms: Part 1: BIIB091 High Dose + Matching Placebo for DRF; Part 1: BIIB091 Low Dose + Matching Placebo for DRF; Part 2: BIIB091 + DRF Low Dose; Part 2: BIIB091 + DRF Standard Dose
Drug: DRF — Administered as specified in the treatment arm.
  Arms: Part 1: DRF + Matching Placebo for BIIB091; Part 2: BIIB091 + DRF Low Dose; Part 2: BIIB091 + DRF Standard Dose; Part 2: DRF + Matching Placebo for BIIB091
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part 1: BIIB091 High Dose + Matching Placebo for DRF; Part 1: BIIB091 Low Dose + Matching Placebo for DRF; Part 1: DRF + Matching Placebo for BIIB091; Part 2: DRF + Matching Placebo for BIIB091

SUMMARY:
In this study, researchers will learn more about a study drug called BIIB091 in participants with MS who may be experiencing relapses. It is a 2-part study.

In Part 1, one set of participants will take either BIIB091 or diroximel fumarate (DRF). In Part 2, a different set of participants will take either a combination of BIIB091 and DRF or DRF alone.

The goal of the study is to learn more about the safety of BIIB091 and to compare the effects of the study drug when taken alone or together with DRF.

The main question researchers are trying to answer are:

* How many participants have new or worsening medical problems (adverse events) after taking BIIB091 or DRF?
* How many new areas of inflammation occur in the brain after treatment with BIIB091 and DRF?

Researchers will use magnetic resonance imaging (MRI) scans to compare images of the brain before and after treatment. They will also explore the effect of BIIB091 and DRF on the heart using electrocardiograms (ECGs).

The study will be done as follows:

* After screening, participants who joined Part 1 will be randomly assigned to receive either a high or low dose of BIIB091, or the standard dose of DRF.
* The results of Part 1 will be used to choose the best dose of BIIB091 to use in Part 2.
* Participants who join Part 2 will be randomly assigned to receive either a standard dose of DRF, a combo of BIIB091 and the standard dose of DRF, or a combo of BIIB91 with a low dose of DRF.
* Neither the researchers nor the participants will know which drug or dose the participants will receive in either part of the study.
* The treatment period will last 48 weeks in each part of the study. Participants will take the drugs by mouth 2 times a day.
* Each part will also have a follow-up safety period that lasts up to 2 weeks.
* In total, participants in each part will have 20 study visits, or more if they have a relapse. The total study duration for participants will be up to 54 weeks.

DETAILED DESCRIPTION:
The primary objectives of this study are to investigate the safety and tolerability of BIIB091 monotherapy in participants with relapsing multiple sclerosis (RMS) in Part 1 and to evaluate the effects of BIIB091 combination therapy with DRF compared with the DRF monotherapy arm on the key MRI measure of active central nervous system (CNS) inflammation in Part 2.

The secondary objectives of Part 1 of the study are to evaluate the effects of BIIB091 monotherapy on the MRI measures of active CNS inflammation and to assess the effect of BIIB091 monotherapy on QTc and other ECG parameters. The secondary objectives of Part 2 are to evaluate the effects of BIIB091 combination therapy with DRF compared with the DRF monotherapy arm on additional MRI measures of active CNS inflammation, the safety and tolerability of BIIB091 combination therapy with DRF in participants with RMS, and the effect of BIIB091 combination therapy with DRF on QTc and other ECG parameters.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of RMS [relapsing-remitting multiple sclerosis (RRMS) or active secondary progressive multiple sclerosis (SPMS)] in accordance with the 2017 Revised McDonald criteria.
2. Time since MS symptom onset is <20 years.
3. Must have expanded disability status scale (EDSS) score of 0 through 5.0 at screening and baseline.
4. Must have at least 1 of the following occurring prior to Baseline (Day 1):

   * ≥2 clinical relapses in the last 24 months (but not within 30 days prior to Baseline [Day 1]) with at least 1 relapse during the last 12 months prior to randomization.
   * ≥1 clinical relapse within the past 24 months (but not within 30 days prior to Baseline [Day 1]) and ≥1 new brain MRI lesion (Gd-positive and/or new or enlarging T2 hyperintense lesion) within the past 12 months prior to randomization. The screening MRI could be used to satisfy this criterion (if needed for inclusion, local reading is required). For new or enlarging T2 hyperintense lesions, the reference scan cannot be >12 months prior to randomization.
   * ≥1 GdE lesion on brain MRI within 6 months prior to randomization.

Key Exclusion Criteria:

1. Diagnosis of primary progressive multiple sclerosis (PPMS) in accordance with the 2017 Revised McDonald criteria.
2. An MS relapse that has occurred within 30 days prior to Baseline (Day 1) or the participant has not stabilized from a previous relapse at the time of screening.
3. History of severe allergic, anaphylactic reactions or hypersensitivity reaction to BIIB091 or DRF, the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study, including the following:

   * Known hypersensitivity to any components of the study treatment
   * Known hypersensitivity to previous fumarate or bruton's tyrosine kinase (BTK) inhibitor treatments
   * History of hypersensitivity to parenteral administration of Gd-based contrast agents
4. Evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within the past 4 weeks prior to Baseline.
5. History of human immunodeficiency virus (HIV) infection or a positive or indeterminate test result at screening for HIV.
6. Current or history of hepatitis C infection regardless of viral load.
7. Current or history of hepatitis B infection.
8. Current enrollment or plan to enroll in any other drug, biological, device, clinical study, or treatment with an investigational drug or approved therapy for investigational use within 90 days prior to randomization or 5 half-lives of the drug or therapy, whichever is longer.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2027-09-07 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) | Day 1 up to Week 50
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product or auxiliary medicinal product, whether or not related to the medicinal (investigational) product or auxiliary medicinal product.
Part 1: Number of Participants With Serious Adverse Events (SAEs) | From signing the informed consent form (ICF) to Week 50
  SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Part 2: Cumulative Number of New T1 Gadolinium-Enhancing (GdE) Lesions | Week 8 to Week 16

SECONDARY OUTCOMES:
Part 1: Cumulative Number of New T1 Gadolinium-Enhancing (GdE) Lesions | Week 8 to Week 16
Part 1: Cumulative Number of New or Enlarging T2 Hyperintense Lesions | Week 8 to Week 16
Part 1: Cumulative Volume of New or Enlarging T2 Hyperintense Lesions | Week 8 to Week 16
Part 1: Mean Change From Baseline in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF), RR, PR, QRS, and QT Intervals | Up to Week 50
Part 1: Number of Participants With Change From Baseline in Heart Rate | Up to Week 50
Part 1: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities | Up to Week 50
Part 2: Cumulative Number of New or Enlarging T2 Hyperintense Lesions | Week 8 to Week 16
Part 2: Cumulative Volume of New or Enlarging T2 Hyperintense Lesions | Week 8 to Week 16
Part 2: Number of Participants With AEs | Day 1 up to Week 50
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product or auxiliary medicinal product, whether or not related to the medicinal (investigational) product or auxiliary medicinal product.
Part 2: Number of Participants With SAEs | From signing of ICF up to Week 50
  SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Part 2: Number of Participants With Change From Baseline in QTcF, RR, PR, QRS, and QT intervals | Up to Week 50
Part 2: Number of Participants With Change From Baseline in Heart Rate | Up to Week 50
Part 2: Number of Participants With ECG Abnormalities as Assessed by 12-Lead ECG Measurements | Up to Week 50

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (77):
- United States (23):
  - HonorHealth Neurology, Scottsdale, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - University of California at Irvine Medical Center, Orange, California
  - University of Colorado School of Medic, Aurora, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - International Neurorehabilitation Institute, Lutherville, Maryland
  - Washington University, St Louis, Missouri
  - Holy Name, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - South Shore Neurologic Associates, P.C., Patchogue, New York
  - Wake Forest University - School of Medicine - Central, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Boster Center for Multiple Sclerosis, Columbus, Ohio
  - Neurology Clinic, PC, Cordova, Tennessee
  - Vanderbilt MS Center, Nashville, Tennessee
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Bulgaria (9):
  - 'MHAT Avis - Medica' OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT 'Sv. Georgi', EAD, Plovdiv
  - MHATNP 'Sv.Naum', EAD, Sofia
  - University First MHAT-Sofia, 'St. Joan Krastitel' EAD, Sofia
  - Acibadem City Clinic Tokuda University Hospital Ead, Sofia
  - DCC Neoclinic EAD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava p.o., Jihlava
  - Fakultni Thomayerova nemocnice, Praha 4-Krc
  - Krajska zdravotni a.s. - Nemocnice Teplice o.z., Teplice
- Germany (6):
  - Studienzentrum fur Neurologie und Psychiatrie, Böblingen, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH- Hohe Warte, Bayreuth, Bavaria
  - Neuropraxis Muenchen Sued, Unterhaching, Bavaria
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - ZNS - Zentrum fuer Neurologisch-Psychiatrische Studien, Siegen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
- Italy (7):
  - I.R.C.C.S. Neuromed-Istituto Neurologico Mediterraneo, Pozzilli, Isernia
  - Fondazione Istituto G.Giglio di Cefalù, Cefalù, Palermo
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
- Poland (14):
  - COPERNICUS Podmiot Leczniczy Sp. z o. o.,, Gdansk
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki
  - Centrum Medyczne Pratia Katowice, Katowice
  - M.A. - LEK A.M.Maciejowscy SC., Katowice
  - Nzoz Novo-Med, Katowice
  - Resmedica Sp.z o.o, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Neurologii K. Selmaj, Lodz
  - Instytut Zdrowia dr Boczarska-Jedynak sp.z.o.o, Sp.K, Oświęcim
  - Med-Polonia Sp. z o.o., Poznan
  - NZOZ 'NEURO-KARD', 'Ilkowski i Partnerzy' Sp. Partn. Lek., Poznan
  - Nzoz Palomed, Rzeszów
  - NeuroProtect Sp. z o.o., Warsaw
  - Wielospecjalistyczne Centrum Medyczne Ibismed, Zabrze
- Caribbean Center for Clinical Research, Guaynabo, San Juan, Puerto Rico
- Romania (3):
  - S.C Neurocity S.R.L, Bucharest
  - Spitalul Universitar de Urgenta Elias, Bucharest
  - S.C Clubul Sanatatii SRL, Campulung Muscel
- Spain (6):
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
- Switzerland (3):
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitaetsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/